CLINICAL TRIAL: NCT02804347
Title: The Effects of Electroconvulsive Therapy (ECT) and/or Intermittent Theta Burst Stimulation (iTBS) on Olfaction and Cognition in Patients With Depression
Brief Title: The Effects of ECT and/or iTBS on Olfaction and Cognition in Patients With Depression
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: Providence Healthcare (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Dr. Roumen Milev, Queen's University
Other Study IDs: 6006093
Record Dates: First submitted 2016-06-02; First posted 2016-06-17 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Depression
Keywords: Olfactory Dysfunction; Electroconvulsive Therapy; Theta Burst Stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient: Patients will be receiving either ECT or iTBS as a depression management. Olfactory functioning will be assessed at pre-treatment and 6 weeks later at post-treatment using Sniffin Sticks. Cognition will also be tested using Cognitive Function Imaging and Battery in the fMRI as well as Cognitive Batteries outside of the scanner at pre-treatment, 6 weeks later at post-treatment, and 3 months after the final treatment session.
  Interventions: Device: Cognitive Function Imaging and Battery; Device: Sniffin Sticks; Other: Cognitive Batteries
- Control: Controls will have their olfactory functioning assessed at baseline and 6 weeks after the baseline assessment using Sniffin Sticks. Cognition will also be tested using Cognitive Function Imaging and Battery in the fMRI as well as Cognitive Batteries outside of the scanner at pre-treatment, 6 weeks later at post-treatment, and 3 months after the final treatment session.
  Interventions: Device: Cognitive Function Imaging and Battery; Device: Sniffin Sticks; Other: Cognitive Batteries

INTERVENTIONS:
Device: Cognitive Function Imaging and Battery — Individuals will be placed in the fMRI scanner and complete the NBACK Cognitive Task
Device: Sniffin Sticks — Using Sniffin Sticks, olfactory functioning will be assessed using three tests: identification, discrimination, and threshold.
Other: Cognitive Batteries — Participants will conduct the following cognitive batteries: DSST, TMT A & B, RAVLT

SUMMARY:
The sense of smell and cognition are known to be closely associated with mood and emotional processes. However, despite the clear links between olfaction and cognitive processes with emotional states, research into the role of olfaction, cognition, and mood disorders has so far yielded variable results. This study proposes to investigate the ability to detect and identify odours and assess cognition in a group of patients with unipolar and bipolar depression prior to and after receiving their scheduled electroconvulsive therapy (ECT) or intermittent theta burst stimulation (iTBS) treatments. Olfaction will be evaluated utilizing standard olfactory testing protocols using commercially available kits. Cognition will be evaluated utilizing standard cognitive test protocols in a functional magnetic resonance imaging protocol. The results will potentially shed light on the link between olfaction, cognition and mood disorders.

DETAILED DESCRIPTION:
The research to date indicates that olfactory sensitivity and cognition are reduced in depressed patients. The data also suggest that higher order cognitive odour evaluation, measured via identification testing, is not altered in depression. Furthermore, research into the effect (if any) of treatment on olfactory performance (sensitivity and identification) has been sparse. Researchers have called for studies that examine olfactory sensitivity prior to psychiatric treatment and post-remission. To the best of our knowledge there has yet to be a study on the effect of electroconvulsive therapy (ECT) or intermittent theta burst stimulation (iTBS) treatments on the olfactory performance of patients with treatment refractory Major Depressive Disorder (MDD) and bipolar depression. ECT has been identified as today's most effective treatment for severe depression due to the remission rates, speed of response, and the completeness of remission. iTBS is a new remittent transcranial magnetic stimulation (rTMS) protocol that has gained more notoriety within the field for the speed of administration, effectiveness of the treatment, and speed of response. Unlike rTMS, TBS mimics the endogenous theta rhythms of the brain, which results in greater potency in inducing long-term potentiation of synaptic connections in the targeted brain regions. iTBS has been shown to be effective in treating mood disturbances, and increasing plasticity and inducing neurogenesis in patients. People with MDD often struggle with cognitive impairments such as decreased executive functioning, attention, concentration, speed of processing, and working memory. The brain areas associated with cognition, such as the prefrontal cortex and hippocampus are negatively affected by depression; studies have shown decreased volume, activity, and disturbed brain connectivity in those two areas. Currently, there is a lack of treatment options for improving cognition in depressed patients. The investigators are focussing on exploring the therapeutic potential of iTBS on cognition.The preliminary evidence from our study will add to scientists' understanding of the short and long term effects of iTBS treatment on the cognitive related areas in the brain through the use of fMRI. The investigators also hope our research will allow psychiatrists to deliver better care to patients with debilitating cognitive impairments associated with depression. Overall, a study examining the olfactory and cognitive performance of patients with treatment resistant MDD and bipolar depression, pre-ECT/iTBS, post-ECT/iTBS, and post-remission would yield valuable insight into the link between olfaction and mood disorders as well as cognition and mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Signed Patient Informed Consent
* Patients with MDD (DSM-IV-TR - criteria used) OR Patients with bipolar depression (DSM-IV-TR - criteria used)
* Males or females over 18 years of age
* In-patients or out-patients currently scheduled to receive ECT or rTMS

Exclusion Criteria:

* Patients suffering from other neurological or endocrine disorders known to affect olfactory functioning.
* Patients suffering from a respiratory tract infection or other respiratory disorder known to affect olfactory functioning at investigator's discretion
* Schizophrenia, Schizoaffective or other Psychotic Disorder
* Patients over 65 years of age
* Patients with significant allergies
* Patients with environmental sensitivities (e.g. perfumes)
* Patients with mechanical obstruction of the nasal passages (e.g. deviated septum)
* Patients with congenital anosmia or other previous primary olfactory dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients receiving iTBS or ECT at Providence Continuing Care Mental Health Services Site and healthy controls recruited from the Kingston Area. Patients may originate from a number of locations and clinics in the area but receive their treatment at Providence Care and have been referred to this location for such. Controls should be age and gender matched to participants and will be recruited from the Kingston region.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Olfactory Function Change using Burghart's Sniffin' Sticks | Baseline and 6 weeks
Cognitive Function Change using NBACK, Shopping List, and Symbol Span Tests | Baseline, 6 weeks, 3 months

SECONDARY OUTCOMES:
Participant's Olfactory Identification using Sniffin' Sticks Identification Test | Baseline and 6 weeks
Participant's Olfactory Threshold using Sniffin' Sticks Threshold Test | Baseline and 6 weeks
Participant's Olfactory Discrimination using Sniffin' Sticks DiscriminationTest | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roumen V Milev, MD FRCPC, Principal Investigator — Queen's University Department of Psychiatry

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ludvigson, H.W., & Rottman, T.R. (1989). Effects of ambient odours of lavender and cloves on cognition, memory, affect, and mood. Chemical Senses, 14(4), 525-536.
- [Background] Albrecht J, Wiesmann M. [The human olfactory system. Anatomy and physiology]. Nervenarzt. 2006 Aug;77(8):931-9. doi: 10.1007/s00115-006-2121-z. German. PMID 16871378
- [Background] Amsterdam JD, Settle RG, Doty RL, Abelman E, Winokur A. Taste and smell perception in depression. Biol Psychiatry. 1987 Dec;22(12):1481-5. doi: 10.1016/0006-3223(87)90108-9. No abstract available. PMID 3676376
- [Background] Austin MP, Mitchell P, Goodwin GM. Cognitive deficits in depression: possible implications for functional neuropathology. Br J Psychiatry. 2001 Mar;178:200-6. doi: 10.1192/bjp.178.3.200. PMID 11230029
- [Background] Berendse HW, Ponsen MM. Detection of preclinical Parkinson's disease along the olfactory trac(t). J Neural Transm Suppl. 2006;(70):321-5. doi: 10.1007/978-3-211-45295-0_48. PMID 17017547
- [Background] Brand G, Millot JL, Henquell D. Complexity of olfactory lateralization processes revealed by functional imaging: a review. Neurosci Biobehav Rev. 2001 Mar;25(2):159-66. doi: 10.1016/s0149-7634(01)00005-7. PMID 11323080
- [Background] Castaneda AE, Tuulio-Henriksson A, Marttunen M, Suvisaari J, Lonnqvist J. A review on cognitive impairments in depressive and anxiety disorders with a focus on young adults. J Affect Disord. 2008 Feb;106(1-2):1-27. doi: 10.1016/j.jad.2007.06.006. Epub 2007 Aug 20. PMID 17707915
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Drevets WC. Functional anatomical abnormalities in limbic and prefrontal cortical structures in major depression. Prog Brain Res. 2000;126:413-31. doi: 10.1016/S0079-6123(00)26027-5. PMID 11105660
- [Background] Frodl T, Meisenzahl EM, Zetzsche T, Born C, Groll C, Jager M, Leinsinger G, Bottlender R, Hahn K, Moller HJ. Hippocampal changes in patients with a first episode of major depression. Am J Psychiatry. 2002 Jul;159(7):1112-8. doi: 10.1176/appi.ajp.159.7.1112. PMID 12091188
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Gentner R, Wankerl K, Reinsberger C, Zeller D, Classen J. Depression of human corticospinal excitability induced by magnetic theta-burst stimulation: evidence of rapid polarity-reversing metaplasticity. Cereb Cortex. 2008 Sep;18(9):2046-53. doi: 10.1093/cercor/bhm239. Epub 2007 Dec 28. PMID 18165282
- [Background] Golinkoff M, Sweeney JA. Cognitive impairments in depression. J Affect Disord. 1989 Sep-Oct;17(2):105-12. doi: 10.1016/0165-0327(89)90032-3. PMID 2527885
- [Background] Gross-Isseroff R, Luca-Haimovici K, Sasson Y, Kindler S, Kotler M, Zohar J. Olfactory sensitivity in major depressive disorder and obsessive compulsive disorder. Biol Psychiatry. 1994 May 15;35(10):798-802. doi: 10.1016/0006-3223(94)91142-8. PMID 8043710
- [Background] Hawkes C. Olfaction in neurodegenerative disorder. Mov Disord. 2003 Apr;18(4):364-72. doi: 10.1002/mds.10379. PMID 12671941
- [Background] Kellner CH, Fink M. The efficacy of ECT and "treatment resistance". J ECT. 2002 Mar;18(1):1-2. doi: 10.1097/00124509-200203000-00001. No abstract available. PMID 11925510
- [Background] Lombion-Pouthier S, Vandel P, Nezelof S, Haffen E, Millot JL. Odor perception in patients with mood disorders. J Affect Disord. 2006 Feb;90(2-3):187-91. doi: 10.1016/j.jad.2005.11.012. Epub 2005 Dec 27. PMID 16376994
- [Background] Martzke JS, Kopala LC, Good KP. Olfactory dysfunction in neuropsychiatric disorders: review and methodological considerations. Biol Psychiatry. 1997 Oct 15;42(8):721-32. doi: 10.1016/s0006-3223(96)00442-8. No abstract available. PMID 9325566
- [Background] Negoias S, Croy I, Gerber J, Puschmann S, Petrowski K, Joraschky P, Hummel T. Reduced olfactory bulb volume and olfactory sensitivity in patients with acute major depression. Neuroscience. 2010 Aug 11;169(1):415-21. doi: 10.1016/j.neuroscience.2010.05.012. Epub 2010 May 13. PMID 20472036
- [Background] Pause BM, Miranda A, Goder R, Aldenhoff JB, Ferstl R. Reduced olfactory performance in patients with major depression. J Psychiatr Res. 2001 Sep-Oct;35(5):271-7. doi: 10.1016/s0022-3956(01)00029-2. PMID 11591429
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Rolls ET, Kringelbach ML, de Araujo IE. Different representations of pleasant and unpleasant odours in the human brain. Eur J Neurosci. 2003 Aug;18(3):695-703. doi: 10.1046/j.1460-9568.2003.02779.x. PMID 12911766
- [Background] Satoh S, Morita N, Matsuzaki I, Konishi T, Nakano T, Minoshita S, Arizono H, Saito S, Ayabe AS. Relationship between odor perception and depression in the Japanese elderly. Psychiatry Clin Neurosci. 1996 Oct;50(5):271-5. doi: 10.1111/j.1440-1819.1996.tb00563.x. PMID 9201790
- [Background] Seo HS, Jeon KJ, Hummel T, Min BC. Influences of olfactory impairment on depression, cognitive performance, and quality of life in Korean elderly. Eur Arch Otorhinolaryngol. 2009 Nov;266(11):1739-45. doi: 10.1007/s00405-009-1001-0. Epub 2009 Jun 2. PMID 19488777
- [Background] Serby M, Larson P, Kalkstein D. Olfactory sense in psychoses. Biol Psychiatry. 1990 Nov 1;28(9):830. doi: 10.1016/0006-3223(90)90520-c. No abstract available. PMID 2257290
- [Background] Small DM, Jones-Gotman M, Zatorre RJ, Petrides M, Evans AC. Flavor processing: more than the sum of its parts. Neuroreport. 1997 Dec 22;8(18):3913-7. doi: 10.1097/00001756-199712220-00014. PMID 9462465
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Steiner JE, Lidar-Lifschitz D, Perl E. Taste and odor: reactivity in depressive disorders, a multidisciplinary approach. Percept Mot Skills. 1993 Dec;77(3 Pt 2):1331-46. doi: 10.2466/pms.1993.77.3f.1331. PMID 8170789
- [Background] Swiecicki L, Zatorski P, Bzinkowska D, Sienkiewicz-Jarosz H, Szyndler J, Scinska A. Gustatory and olfactory function in patients with unipolar and bipolar depression. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Aug 1;33(5):827-34. doi: 10.1016/j.pnpbp.2009.03.030. Epub 2009 Apr 5. PMID 19345708
- [Background] Van Toller S, Reed MK. Brain electrical activity topographical maps produced in response to olfactory and chemosensory stimulation. Psychiatry Res. 1989 Sep;29(3):429-30. doi: 10.1016/0165-1781(89)90112-1. No abstract available. PMID 2608810
- [Background] Warner MD, Peabody CA, Csernansky JG. Olfactory functioning in schizophrenia and depression. Biol Psychiatry. 1990 Feb 15;27(4):457-8. doi: 10.1016/0006-3223(90)90557-i. No abstract available. PMID 2178695
- [Background] Weismann M, Yousry I, Heuberger E, Nolte A, Ilmberger J, Kobal G, Yousry TA, Kettenmann B, Naidich TP. Functional magnetic resonance imaging of human olfaction. Neuroimaging Clin N Am. 2001 May;11(2):237-50, viii. PMID 11489737
- [Background] Wiesmann M, Kopietz R, Albrecht J, Linn J, Reime U, Kara E, Pollatos O, Sakar V, Anzinger A, Fesl G, Bruckmann H, Kobal G, Stephan T. Eye closure in darkness animates olfactory and gustatory cortical areas. Neuroimage. 2006 Aug 1;32(1):293-300. doi: 10.1016/j.neuroimage.2006.03.022. Epub 2006 May 2. PMID 16631383